CLINICAL TRIAL: NCT00614731
Title: Responses to Immunization With Keyhole Limpet Hemocyanin Administered by Scarification and the Intradermal Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis and Vaccinia Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DAIT ADVN KLH 07; Contract No. HHSN266200400029C
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Atopic Dermatitis
Keywords: Keyhole Limpet Hemocyanin; KLH; atopic dermatitis; IgG antibodies; scarification
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ID immunizations (100 mcg) (Experimental): Participants will receive a total of two 100 mcg intradermal (ID) KLH carrier-protein immunizations with 1 mg/ml KLH per immunization. Immunizations will be given 21 days apart at Visits 5 and 6.
  Interventions: Biological: KLH carrier-protein
- Scarification by 3 jabs (Experimental): Participants will receive two scarification immunizations by 3 jabs containing 20 mg/ml of KLH carrier-protein. The immunizations will occur 21 days apart at Visits 5 and 6.
  Interventions: Biological: KLH carrier-protein
- ID immunizations (250 mcg) (Experimental): Enrollment will begin after the safety data for Groups 1A and 2A have been reviewed. Participants in this group will receive two 250 mcg ID KLH vaccinations containing 10 mg/ml of KLH carrier-protein. Immunizations will occur 21 days apart at Visits 5 and 6.
  Interventions: Biological: KLH carrier-protein
- Scarification by 15 jabs (Experimental): Enrollment will begin after the safety data from groups 1A and 2A has been examined. Participants in this group will receive a total of two scarification immunizations by 5 needles used to administer 15 jabs, each containing, 20 mg/ml of KLH carrier-protein. Immunizations will occur 21 days apart at Visits 5 and 6.
  Interventions: Biological: KLH carrier-protein

INTERVENTIONS:
Biological: KLH carrier-protein — KLH carrier-protein vaccination containing no other protein or antibodies
  Other Names: Immucothel; Vacmune

SUMMARY:
Atopic dermatitis (AD) is a skin disorder in which people often have swelling and skin infections. People with this disease cannot receive the smallpox vaccine because it could cause them to have a fatal reaction known as eczema vaccinatum (EV). Keyhole limpet hemocyanin (KLH) is a protein that can be used to deliver vaccines to the body. The purpose of this study is to determine a baseline immune reaction to KLH in people without AD. Once this has been established, other studies can be designed to determine whether KLH can be used to give vaccines to people with AD.

DETAILED DESCRIPTION:
AD is characterized by skin inflammation and recurrent skin infections. In addition, people with AD may have a severe and sometimes fatal reaction to the smallpox vaccine called EV. KLH is a carrier protein that can be used to deliver antibodies to the body. However KLH itself, may cause an immune response. The purpose of this study is to determine the body's reaction to pure KLH in people without AD. This will be used to establish a baseline immune response and may be compared to the immune response in people with AD during future studies.

This study will last 8 weeks and will have 11 study visits. Participants in this study will be randomly assigned to 1 of 4 groups. All participants will receive their immunizations at Visits 5 and 6. Participants in Group 1A will receive 2 immunizations each with 100 mcg of KLH each. Participants in Group 2A will receive 2 immunizations through scarification (a shallow cut in the skin) with jabs, each containing 20 mg/mL of KLH. Adverse reactions will be monitored after each immunization. Once safety data from these 2 groups have been reviewed, the next 2 groups will be enrolled. Participants in Group 1B will receive 2 immunizations each with 250 mcg of KLH each. Participants in Group 2B will receive 2 immunizations through scarification with 15 jabs, each containing 20mg/mL of KLH. Other study visits will include allergy testing and blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and nonatopic as defined by the ADVN Standard Diagnostic Criteria
* Willing to use appropriate forms of contraception

Exclusion Criteria:

* Active bacterial, viral, or fungal infection within 30 days prior to study entry
* Immunodeficiency
* Received Use of systemic corticosteroids, antibiotics, antivirals, anti-inflammatory biologics (e.g., alefacept, etanercept), calcineurin inhibitors, oral immunosuppressive agents, anxiolytic agents, antidepressants, or cancer chemotherapy within 30 days prior to KLH administration
* Use of topical corticosteroids, antibiotics, antivirals, immune enhancers, or calcineurin inhibitors within 7 days prior to study entry
* Allergy to shellfish
* Vaccination within 30 days prior to entering the study
* Skin rash
* Participation in a clinical trial within 4 weeks of study entry
* Positive response to DTH test prior to administration of KLH
* Previous exposure to KLH or products containing KLH
* Allergic or hypersensitivity to KLH
* Any condition that, in the opinion of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in anti-KLH IgG antibody response to two vaccinations of KLH in nonatopic participants | At baseline and Day 47
Safety of administering KLH by scarification route as measured by proportion of subjects with any treatment-emergent abnormalities in vital signs (body temperature, heart rate, respirations, and blood pressure) and liver function | Throughout study

SECONDARY OUTCOMES:
Change in anti-KLH antibody responses in IgG subclasses 1 to 4, IgA, IgM, and IgE. | At baseline and Day 47
Incidence of all adverse events (AEs) | Throughout study
Change in diameter of delayed type hypersensitivity (DTH) responses to KLH | At Day 2 and 49
Induction of a T cell response as measured by a change from negative (smaller than 5 mm) to positive (5 mm or larger) DTH reaction. | At Days 2 and 49
Presence or absence of antibody response as measured by whether or not there is a greater than 2 fold increase in antibody (IgG, IgA, IgM, IgE) titers to two administrations of KLH. | At Days 0 and 47
Changes pre- versus post-administration of KLH in quantitative levels of clinical labs (CBC, liver function [AST, ALT], renal function [creatinine, BUN]) | At Days 0 and 47
Changes pre- versus post-administration of KLH in quantitative levels of vital signs (body temperature, heart rate, respirations, blood pressure) | At Days 0 and 47

CONTACTS AND LOCATIONS:
Overall Officials: Henry Milgrom, M.D., Principal Investigator — National Jewish Health; Donald Y Leung, M.D., Ph.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Milgrom H, Kesler K, Byron M, Harbeck R, Holliday R, Leung DY. Response to cutaneous immunization with low-molecular-weight subunit keyhole limpet hemocyanin. Int Arch Allergy Immunol. 2012;157(3):269-74. doi: 10.1159/000328784. Epub 2011 Oct 28. PMID 22042247
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY3 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY3 — ImmPort study identifier is SDY3.
- Available data/document: Study Protocol: SDY3 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY3 — ImmPort study identifier is SDY3.
- Available data/document: Study design, -schedule of events, -demographics, -adverse events, -interventions, -files: SDY3 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY3 — ImmPort study identifier is SDY3.